CLINICAL TRIAL: NCT05751460
Title: Translation and Validation of Pelvic Girdle Questionnaire in Urdu Language
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Faiza Kalsoom
Record Dates: First submitted 2022-10-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Straight leg raise — Diagnostic test, tool for *g*
  Other Names: Pelvic girdle questionnaire

SUMMARY:
Urdu version of pelvic girdle questionnaire was drafted, tested for its reliability and validity on patients with pelvic girdle pain. Urdu version was linguistically acceptable and accurate for pregnant and post partum females with pelvic girdle pain. The result seems comparable to all the other versions and especially with original Norwegian version. This instrument is understandable and easy to find disability during pregnancy and post partum duration. It showed a good content, construct and convergent validity also present high internal consistency and test retest reliability.

DETAILED DESCRIPTION:
The Pelvic Girdle Questionnaire is the only specific instrument designed to evaluate pain and activity limitations in pregnant or postpartum women with pelvic girdle pain. This study aimed to translate the Pelvic girdle questionnaire in Urdu language for Pakistani female patients and to verify the validation of the psychometric items of the Pelvic girdle questionnaire in population of Pakistan. The purpose of this study was to translate the Pelvic Girdle Questionnaire into Urdu and find out cross-culture validity and reliability of Urdu Pelvic girdle questionnaire among pregnant and postpartum females. A cultural adaptation and translation study was performing according to international guidelines. Study was conducted at different hospital settings. Pre test was conducted among 16 females during pregnancy & post-partum.

Key words: Disability Evaluation, Female, Urdu, Pelvic Girdle Pain and physiopathology, Pregnancy, Surveys and Questionnaires, Translation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Only Females
* Able to read Urdu Language
* Pregnant women (gestational week 30-38)
* Postpartum women (given birth less than one year earlier)

Exclusion Criteria:

* Any neurological diseases (reflex changes & loss of sensation)
* Unstable medical conditions leading to fatigue
* Those that have prolapse or severe urinary disease
* Previous surgery on pelvis, lower limb or spine
* Cannot Understand Urdu
* Difficulty in understanding the Pelvic girdle questionnaire

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female pregnant and post partum with pelvic girdle pain
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Content validity | "through study completion, an average of 1 year"
  Content validity score measured by content validity index. Assessment of 25 items by Clinician and native speaker experts rate all the items and all the value are above 0.70.Lower value was 0.92 and the highest value is 1 which is maximum value. Maximum score is given to 4, 5, 6,10,11,12,17,18,22 and 24 by experts (medical specialist and native speakers).

SECONDARY OUTCOMES:
Internal consistency: | "upto two weeks"
  Cronbach's alpha was used for reliability. The reliability and internal consistency of PGQ for PGP patients Cronbach's alpha in week one and week two is 0.977 and 0.976 respectively. The value of α for activity subscale (1-20) is 0.986 and symptom subscale (21- 25) is 0.970.

OTHER OUTCOMES:
Convergent validity | "through study completion, an average of 1 year"
  The value of Pearson correlation coefficient for Pelvic girdle questionnaire with Ostwestry disability index is 0.840 and NRS is 0.772.For the calculation of construct validity of PGQ we used Pearson's correlation coefficient with 5% significance. The correlation between week 1 and week 2 for each item of PGQ scale was ranging from 0.871-0.990. . We compared PGQ with ODI scale and Numeric rating pain scale. The construct validity of PGQ was measured by confidence interval 95% and level of significance at 5%.
Test Retest reliability: | "through study completion, an average of 1 year"
  The tool reliability analyzes by ICC. The value of Intra class correlation for PGQ is 0.979 with 95 % of confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Abdul Hameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Faiza Kalsoom, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cong H, Liu H, Sun Y, Gao J, Liu J, Ma L, Stuge B, Chen L. Cross-cultural adaptation, reliability, and validity of a Chinese version of the pelvic girdle questionnaire. BMC Pregnancy Childbirth. 2021 Jun 30;21(1):470. doi: 10.1186/s12884-021-03962-8. PMID 34193061
- [Background] Sakamoto A, Hoshi K, Gamada K. Transcultural Reliability and Validity of the Japanese-Language Version of the Pelvic Girdle Questionnaire. J Manipulative Physiol Ther. 2020 Jan;43(1):68-77. doi: 10.1016/j.jmpt.2018.11.019. Epub 2020 Feb 13. PMID 32061416
- [Background] Acharya RS, Tveter AT, Grotle M, Khadgi B, Koju R, Eberhard-Gran M, Stuge B. Cross-Cultural Adaptation and Validation of the Nepali Version of the Pelvic Girdle Questionnaire. J Manipulative Physiol Ther. 2020 Mar-Apr;43(3):257-265. doi: 10.1016/j.jmpt.2019.04.009. Epub 2020 Jul 29. PMID 32739042
- [Background] Munisamy A, Sahid, Sheerad Hussin, Muhammad. Content Validation and Content Validity Index Calculation of B40 Household's Financial Literacy. Turkish Online Journal of Qualitative Inquiry. 202112(8).
- [Background] Dunn G, Egger MJ, Shaw JM, Yang J, Bardsley T, Powers E, Nygaard IE. Trajectories of lower back, upper back, and pelvic girdle pain during pregnancy and early postpartum in primiparous women. Womens Health (Lond). 2019 Jan-Dec;15:1745506519842757. doi: 10.1177/1745506519842757. PMID 30991911
- [Background] Gutke A, Stuge B, Elden H, Sandell C, Asplin G, Fagevik Olsen M. The Swedish version of the pelvic girdle questionnaire, cross-cultural adaptation and validation. Disabil Rehabil. 2020 Apr;42(7):1013-1020. doi: 10.1080/09638288.2018.1515991. Epub 2019 Feb 1. PMID 30707631
- [Background] Rashidi Fakari F, Kariman N, Ozgoli G, Ghare Naz MS, Ghasemi V, Rashidi Fakari F, Ebadi A. Iranian version of Pelvic Girdle Questionnaire: Psychometric properties and cultural adaptation. J Res Med Sci. 2019 May 22;24:43. doi: 10.4103/jrms.JRMS_391_18. eCollection 2019. PMID 31160910
- [Background] Fagundes FML, Cabral CMN. Cross-cultural adaptation of the Pelvic Girdle Questionnaire (PGQ) into Brazilian Portuguese and clinimetric testing of the PGQ and Roland Morris questionnaire in pregnancy pelvic pain. Braz J Phys Ther. 2019 Mar-Apr;23(2):132-139. doi: 10.1016/j.bjpt.2018.11.003. Epub 2018 Nov 17. PMID 30501939
- [Background] Starzec M, Truszczynska-Baszak A, Stuge B, Tarnowski A, Rongies W. Cross-cultural Adaptation of the Pelvic Girdle Questionnaire for the Polish Population. J Manipulative Physiol Ther. 2018 Oct;41(8):698-703. doi: 10.1016/j.jmpt.2018.04.002. Epub 2018 Dec 26. PMID 30594333
- [Background] Girard MP, O'Shaughnessy J, Doucet C, Lardon E, Stuge B, Ruchat SM, Descarreaux M. Validation of the French-Canadian Pelvic Girdle Questionnaire. J Manipulative Physiol Ther. 2018 Mar-Apr;41(3):234-241. doi: 10.1016/j.jmpt.2018.01.001. Epub 2018 Feb 15. PMID 29456093